CLINICAL TRIAL: NCT00172770
Title: The Establishment of the Early Intervention Program for Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Other Study IDs: 93621700617; DOH93-TD-M-113-032
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Schizophrenia is a severe mental illness, which has a prodromal phase of 1-2 years prior to the onset of the illness. During the prodromal phase, patients might show maladaptation and/or poor social functioning. However, these early symptom of schizophrenia might be overlooked by patients and their families. At that period, patients might strive to improve their social interactions and social functioning. However, the efforts might further create their stress level on everyday life, which can actually accelerate the illness onset of schizophrenia. In other words, the efforts would worsen the pathophysiologic changes in the brain, which can result in the positive symptoms of schizophrenia.

Previous researches found that the critical period for treatment of schizophrenia is the early phase of illness onset, especially the first two or three years. Delay treatment would worsen the illness. To this extent, early treatment would bring to a better prognosis as well as minimize the costs of individuals, families and society. In other words, early interventions not only can prevent relapse, it also can benefit patients' psychosocial adjustments. However, researches found that the average duration of untreated psychosis is 25.2 months in Taiwan, which indicates the phenomena of delay treatment and this trend might result in missing the critical treatment period.

This is a two years study aiming to establish an early intervention program for patients with schizophrenia. In the first year, it aims to understand the phenomena of psychiatric care services utilization for patients with schizophrenia, special emphasis will be on the delay treatment and pluralistic health seeking process. In the second year, it aims to establish an early intervention program. The results of this research would contribute to in-service trainings, service providing, and policy making of psychiatric services.

ELIGIBILITY:
Inclusion Criteria:

* patients with schizophrenia
* capable to express in Chinese
* willing to cooperate with

Exclusion Criteria:

* patients with schizophrenia but not willing to cooperate with

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Chuan Hsiung, Ph.D, Study Chair — Department of Nursing, National Taiwan University
Locations (1):
- Ping-Chuan,Hsiung, Taipei, Taiwan